CLINICAL TRIAL: NCT05293093
Title: Clinical Evaluation and Effectiveness of the Adapted Wheelchair Skills Training Program in People With Complex Movement Disorders
Brief Title: Effectiveness of the Wheelchair Skills Training Program in People With Complex Movement Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Elegast Monbaliu, Prof., KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S65462
Record Dates: First submitted 2022-03-02; First posted 2022-03-24 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: A one-group pretest-posttest design study will be conducted, consisting of three phases (3- or 5-week baseline phase, 4-week training phase, 4-week retention phase) and four wheelchair skill capacity assessment points (T0: baseline; T1: pre-intervention; T2: post-intervention; T3: retention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wheelchair Skills Training Program intervention study (Experimental): A one-group pretest-posttest design study will be conducted, consisting of three phases (3- or 5-week baseline phase, 4-week training phase, 4-week retention phase)
  Interventions: Other: Wheelchair Skills Training Program

INTERVENTIONS:
Other: Wheelchair Skills Training Program — a standardized training method for users of manual and powered wheelchairs and it combines evidence on motor-skills learning with evidence on how to perform specific wheelchair skills. A recent systematic review and meta-analysis provided evidence that WSTP is a safe and effective intervention that has a clinically meaningful effect on powered wheelchair skill capacity, in particular for new wheelchair users. The WSTP has shown to be effective in several wheelchair-dependent populations and promising to be used in people with complex movement disorders. Yet, adaptation to the specific needs and capabilities of individuals with complex movement disorders is necessary as it has not been assessed in this population. During the 4-week training phase, the participants will receive 3 training sessions per week of 45 minutes, including exercises as described in the Wheelchair Skill Training Program Version 5.1.2

SUMMARY:
The overall goal of this project is to increase independent mobility in populations with complex movement disorders, such as severe cerebral palsy, by adapting The Wheelchair Skills Training Program (WSTP) to the needs and capabilities of this population. The primary objective is to evaluate the clinical effectiveness of an adapted Wheelchair Skills Training Program tailored for children with complex movement disorders and its impact on wheelchair mobility skills. Secondary objectives are to evaluate the clinical effectiveness of an adapted Wheelchair Skills Training Program tailored for children with complex movement disorders, and its impact on stress, fatigue, and symptoms of the movement disorder, and to evaluate the clinical effectiveness of an adapted Wheelchair Skills Training Program tailored for children with complex movement disorders, and its impact on participation. The investigators hypothesize an improvement in wheelchair skill capacity and performance post-intervention compared to pre-intervention. In addition, the investigators hypothesize that the levels of stress and fatigue are in the general low to moderate throughout the training sessions. However, the investigators also expect that higher levels of (perceived) stress and fatigue negatively impact task performance and provoke the symptoms of the movement disorder. The investigators hypothesize that participation will improve post-intervention compared to pre-intervention.

DETAILED DESCRIPTION:
Powered wheelchair training for individuals with complex movement disorders, such as severe cerebral palsy, is challenging for healthcare providers, funders, and patients: it is highly dependent on the expertise of training staff (e.g., physical and occupational therapists), time-consuming for staff and patients, and therefore costly for providers. Poor personalisation of current training protocols leads to insufficient clinical outcomes. The overall goal of this project is to increase independent mobility in populations with complex movement disorders, such as severe cerebral palsy, by adapting The Wheelchair Skills Training Program (WSTP) to the needs and capabilities of this population.

This study focuses on the effectiveness and clinical evaluation of the Wheelchair Skills Training Program (WSTP), adapted for children with complex movement disorders. Despite the proven effectiveness of the WSTP in other wheelchair-dependent populations, it warrants cautious implementation in clinical and educational settings within our target population of children with Dyskinetic and Spastic CP (GMFCS III- V). The project contains three study objectives. In the first objective, the effectiveness of a powered-wheelchair skill training program (WSTP) tailored for children with complex movement disorders on wheelchair mobility skills will be assessed. In the second study objective, the impact of a powered-wheelchair training session on measures as stress, motivation and fatigue will be evaluated. In the third study objective, the effect on everyday participation and quality of life will be assessed.

The primary endpoint is the wheelchair mobility skill performance, assessed using the Wheelchair Skills Test (WST). This is an objective test of a set of wheelchair skills. It is proven to be a reliable and valid assessment tool and is used in a number of studies as an outcome measure for (powered) wheelchair skills capacity. The main advantage of the WST is that the tester can see how the wheelchair user carries out the skill, permitting problems due to the wheelchair or the technique used to be identified and addressed.

Although WST capacity measures have been found to be sensitive to changes due to training, other measures will also be used to identify training effects on wheelchair mobility skills as recommended. The Wheelchair Skills Test - Questionnaire (WST-Q) will be used as it allows to assess performance as well as capacity and that in subject's own setting which together with WST is recommended for a comprehensive assessment.

Secondary endpoints include measures such as heart rate variability to explore the impact of stress and fatigue on task performance. Emotion Faros 360° devices will be used. Secondary endpoints also include measures of establishing the relationship of the intervention program with the subject's perceived exertion, Intrinsic Motivation Inventory questionnaire, participation by Canadian Occupational Performance Measure (COPM), and quality of life via the CP-QoL.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Cerebral Palsy
* classified as level III-V on the Gross Motor Function Classification System
* classified as level III-V on the Manual Ability Classification System
* must be able to understand mobility training instructions
* must be currently using a powered wheelchair

Exclusion Criteria:

* underwent surgery of neurological nature less than 12 months prior to the start of the study
* known diagnosis of autism spectrum disorder
* history of traumatic brain injury since diagnosis of cerebral palsy
* history of epilepsy

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Wheelchair mobility skill performance at Post-Intervention assessed by the Wheelchair Skills Test (WST). | 4-week Wheelchair Skills Training Program intervention period (starting from the end of the baseline period)
  The change from Baseline Wheelchair mobility skill performance at Post-Intervention will be assessed using the Wheelchair Skills Test (WST). This is an objective test of a set of wheelchair skill tasks, where wheelchair mobility skill performance is scored as a percentage between 0-100% (higher scores indicate a better wheelchair mobility skill performance).
Change from Post-Intervention Wheelchair mobility skill performance after a 4-week retention period assessed by the Wheelchair Skills Test (WST). | 4-week retention period (starting from the end of the intervention period)
  The change from Post-Intervention Wheelchair mobility skill performance after a 4-week retention period will be assessed using the Wheelchair Skills Test (WST). This is an objective test of a set of wheelchair skill tasks, where wheelchair mobility skill performance is scored as a percentage between 0-100% (higher scores indicate a better wheelchair mobility skill performance).

SECONDARY OUTCOMES:
Monitoring of Heart Rate Variability measured by the eMotion Faros 360° Heart rate variability Sensor during the experiments. | 11-13 weeks (starting from the beginning of the baseline period until the end of the retention period)
  Heart rate variability (HRV) is the fluctuation in the time intervals (in ms) between adjacent heartbeats. The heart rate variability of the participants will be monitored during the training sessions in the intervention period. HRV indexes neurocardiac function and is generated by heart-brain interactions and dynamic non-linear autonomic nervous system processes. HRV is an emergent property of interdependent regulatory systems which operate on different time scales to help persons to adapt to environmental and psychological challenges, and is used as an indicator for stress.
Change in Baseline Participation goals assessed by the Canadian Occupational Performance Measure assessment tool at Post-intervention | 4-week intervention period (starting from the end of the baseline period)
  The Canadian Occupational Performance Measure assessment tool identifies three participation goals per participant. Each identified goal is scored on 'importance', 'execution' and 'satisfaction' using a 1 - 10 scale (higher scores indicate a better outcome)
Change in Post-intervention Participation goals assessed by the Canadian Occupational Performance Measure assessment tool after a 4-week retention period | 4-week retention period (starting from the end of the intervention period)
  The Canadian Occupational Performance Measure assessment tool identifies three participation goals per participant. Each identified goal is scored on 'importance', 'execution' and 'satisfaction' using a 1 - 10 scale (higher scores indicate a better outcome)
Change from Baseline Quality of Life assessed by the Cerebral Palsy Quality of Life Questionnaire for Children (CP QOL-Child) at Post-intervention | 4-week intervention period (starting from the end of the baseline period)
  The Cerebral Palsy Quality of Life Questionnaire for Children (CP QOL-Child) comprises 66 items. Items are transformed to a scale with a possible range of 0-100 (higher scores indicate a better outcome).
Change from Baseline Quality of Life assessed by the Cerebral Palsy Quality of Life Questionnaire for Adolescents (CP QOL-Teen) at Post-intervention | 4-week intervention period (starting from the end of the baseline period)
  The Cerebral Palsy Quality of Life Questionnaire for Adolescents (CP QOL-Teen) comprises 88 items. Items are transformed to a scale with a possible range of 0-100 (higher scores indicate a better outcome).
Change from Post-intervention Quality of Life assessed by the Cerebral Palsy Quality of Life Questionnaire for Children (CP QOL-Child) after a 4-week retention period | 4-week retention period (starting from the end of the intervention period)
  The Cerebral Palsy Quality of Life Questionnaire for Children (CP QOL-Child) comprises 66 items. Items are transformed to a scale with a possible range of 0-100 (higher scores indicate a better outcome).
Change from Post-intervention Quality of Life assessed by the Cerebral Palsy Quality of Life Questionnaire for Adolescents (CP QOL-Teen) after a 4-week retention period | 4-week retention period (starting from the end of the intervention period)
  The Cerebral Palsy Quality of Life Questionnaire for Adolescents (CP QOL-Teen) comprises 88 items. Items are transformed to a scale with a possible range of 0-100 (higher scores indicate a better outcome).
Change in Baseline Motivation assessed by the Intrinsic Motivation Inventory questionnaire at Post-intervention | 4-week intervention period (starting from the end of the baseline period)
  The Intrinsic Motivation Inventory (IMI) is a multidimensional measurement device intended to assess participants' subjective experience related to a target activity. The instrument assesses participants' interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, relatedness, and perceived choice while performing a given activity, thus yielding seven subscale scores. The questionnaire used in the study comprises 14 items (two items per subscale) transformed to a score with a possible range of 0-14 (higher scores indicate a better outcome).
Change from Baseline Wheelchair mobility skill performance at Post-Intervention assessed by the Wheelchair Skills Test-Questionnaire (WST-Q). | 4-week intervention period (starting from the end of the baseline period)
  The change from Baseline Wheelchair mobility skill performance at Post-Intervention will be assessed using the Wheelchair Skills Test-Questionnaire (WST-Q). This questionnaire evaluates the (perceived) capacity and performance of a set of wheelchair skill tasks, where wheelchair mobility skill performance is scored as a percentage between 0-100% (higher scores indicate a better wheelchair mobility skill performance).
Change from Post-Intervention Wheelchair mobility skill performance after a 4-week retention period assessed by the Wheelchair Skills Test-Questionnaire (WST-Q). | 4-week retention period (starting from the end of the intervention period)
  The change from Post-Intervention Wheelchair mobility skill performance after a 4-week retention period will be assessed using the Wheelchair Skills Test-Questionnaire (WST-Q). This questionnaire evaluates the (perceived) capacity and performance of a set of wheelchair skill tasks, where wheelchair mobility skill performance is scored as a percentage between 0-100% (higher scores indicate a better wheelchair mobility skill performance).

CONTACTS AND LOCATIONS:
Overall Officials: Elegast Monbaliu, PhD, Principal Investigator — KU Leuven Department of Rehabilitation Sciences, Campus Bruges
Locations (1):
- KU Leuven Department of Rehabilitation Sciences, Campus Bruges, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No